CLINICAL TRIAL: NCT01713413
Title: Effects of an Oxymizer Versus Conventional Nasal Cannula on Endurance Time in Patients With Chronic Obstructive Pulmonary Disease IV (COPD) or Interstitial Lung Disease (ILD)
Brief Title: Effects of an Oxymizer on Endurance Time in Patients With Chronic Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician (department of pneumology), Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OXYM2012
Record Dates: First submitted 2012-02-24; First posted 2012-10-24 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: COPD; Interstitial Lung Disease
Keywords: Oxymizer; endurance time; exercise test; nasal cannula; COPD; ILD; oxygenation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxymizer (Active Comparator): Using first the Oxymizer and 24 h later the conventional nasal cannula.
  Interventions: Device: Oxymizer
- nasal cannula (Active Comparator): Using first the conventional nasal cannula and 24 h later the Oxymizer
  Interventions: Device: conventional nasal cannula

INTERVENTIONS:
Device: Oxymizer — Using first the Oxymizer and 24 h later the conventional nasal cannula.
  Arms: Oxymizer
Device: conventional nasal cannula — Using first the conventional nasal cannula and 24h later the Oxymizer
  Arms: nasal cannula

SUMMARY:
The Oxymizer pendant® is a special oxygen cannula that can be used to supply high flow long term oxygen therapy. It is compatible with a wide variety of oxygen sources. In a reservoir, the Oxymizer® stores pure oxygen so that the concentration of inhaled oxygen is increased.

The aim of this study is to investigate the potential benefit of the Oxymizer® with regard to the blood oxygenation during exercise testing. Given that the "endurance time" is very sensitive for little changes in exercise capacity, this test will be used to show the difference between the Oxymizer® and a conventional nasal cannula regarding exercise duration at 70% of peak Watt and oxygenation.

The tests will be accompanied by blood gas analysis, partial pressure of carbon dioxide and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* COPD IV
* interstitial lung disease
* long-term oxygen therapy with oxygen flow rate >= 2 L/min

Exclusion Criteria:

* acute cardial decompensation
* usual kontraindication for exposure test (higher-grad Hypertension (arterial and pulmonal), cardiac valve vitien, instabile angina pectoris, cardiac arrhythmia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Difference between Endurance time with Oxymizer and conventional nasal cannula | From starting until stopping cycling, up to 60 minutes

SECONDARY OUTCOMES:
Difference in oxygen saturation with Oxymizer and with conventional nasal cannula | stopping cycling, up to 60 minutes
Difference in PaCO2 with Oxymizer and with conventional nasal cannula | Stopping cycling, up to 60 minutes
  measured by Sentec device

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Berchtesgadener Land, Berchtesgaden, Bavaria, Germany